CLINICAL TRIAL: NCT01708369
Title: Inhibition of Carboxylesterase Metabolism by Ethanol
Brief Title: Alcohol Inhibits Drug Metabolism by Carboxylesterases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Principal Investigator, Robbie Parker, Professor, University of Tennessee
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: R15GM096074 (NIH)
Record Dates: First submitted 2012-10-13; First posted 2012-10-16 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Drug Interactions
Keywords: human carboxylesterase-1; human carboxylesterase-2; alcohol; pharmacokinetics
MeSH Terms: interventions — Ethanol; Oseltamivir; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Oseltamivir & Placebo (Active Comparator): Oseltamivir 150 mg orally will be administered 15 minutes after subjects consume orange juice
  Interventions: Drug: Placebo; Drug: Oseltamivir
- Oseltamivir & Ethanol (Experimental): Oseltamivir 150 mg and ethanol targeted to blood alcohol concentration 0.08 g/dl
  Interventions: Drug: Ethanol; Drug: Oseltamivir
- Aspirin & Placebo (Active Comparator): Aspirin 650 mg orally will be administered 15 minutes after subjects consume orange juice
  Interventions: Drug: Placebo; Drug: Aspirin
- Aspirin & Ethanol (Experimental): Aspirin 650 mg and ethanol targeted to blood alcohol concentration 0.08 g/dl
  Interventions: Drug: Ethanol; Drug: Aspirin

INTERVENTIONS:
Drug: Placebo — Orange juice administered 15 minutes before subjects take oseltamivir or aspirin
  Other Names: Tropicana orange juice
  Arms: Aspirin & Placebo; Oseltamivir & Placebo
Drug: Ethanol — Ethanol will be mixed with orange juice and subjects will drink the mixture 15 minutes before receiving oseltamivir or aspirin
  Other Names: Ethanol plus Tropicana orange juice
  Arms: Aspirin & Ethanol; Oseltamivir & Ethanol
Drug: Oseltamivir — Oseltamivir 150 mg orally
  Other Names: Tamiflu
  Arms: Oseltamivir & Ethanol; Oseltamivir & Placebo
Drug: Aspirin — Aspirin 650 mg orally will be given
  Arms: Aspirin & Ethanol; Aspirin & Placebo

SUMMARY:
The purpose of this study is to determine if alcohol is able the affect the body's ability to eliminate two commonly used medication, oseltamivir and aspirin. We hypothesize that drinking alcohol may reduce the body's ability to break down these two medications along with many others.This could affect the amount of drug in the blood which could impact how well these drugs work and whether patients have side effects.

DETAILED DESCRIPTION:
Carboxylesterases are enzymes that metabolize a growing number of commonly used medications. In humans, two carboxylesterases, carboxylesterase-1 (hCE1) and carboxylesterase-2 (hCE2), found primarily in the liver and intestine respectively, play an important role in the biotransformation of numerous classes of commonly used drugs containing ester groups including ACE inhibitors, anticancer agents, opiate analgesics, HMG-CoA reductase inhibitors (statins), CNS stimulants, antiviral medications, and antiplatelet agents.

Factors affecting the activity of carboxylesterases would be expected to markedly alter the pharmacokinetics and clinical effects of substrate drugs. One key factor that could affect catalytic activity is drug interactions that inhibit carboxylesterase function. The importance of inhibition of drug metabolism in medication safety and efficacy is well established for drugs that undergo metabolism by cytochrome P450 enzymes. In distinct contrast, little is known about the potential for carboxylesterases to serve as a target for metabolic inhibition mediated by drug interactions.

It is well established that ethanol is an inhibitor of cocaine metabolism, a drug that is eliminated by carboxylesterase hydrolysis. We propose that the ethanol-mediated inhibition of carboxylesterases activity demonstrated with cocaine metabolism will occur with other substrate drugs. This has widespread implications because of the large number of drugs that are carboxylesterase substrates. In the United States, over 100 million people consume ethanol making co-ingestion with carboxylesterase substrate drugs a common occurrence. We believe that this is a prevalent drug interaction that is largely overlooked and has not been systematically evaluated, but may importantly affect the disposition, safety, and efficacy of these medications. To address this gap, we will evaluate the effect of ethanol on the disposition of oseltamivir, an hCE1 substrate, and aspirin, an hCE2 substrate, in humans.

Normal healthy volunteers will report to the University of Tennessee Health Science Center Clinical Research Center (CRC) for a 10 hour stay on four separate days and receive each of the following treatments in random order:

1. Oseltamivir (Tamiflu®) 150 mg. Subjects will drink orange juice (about 10 ounces although the amount may vary slightly based on weight) over 15 minutes. Fifteen minutes after drinking the orange juice, subjects will receive two (2) 75 mg capsules of oseltamivir with 5 ounces of water. Blood samples (1 teaspoonful) to determine the amount of oseltamivir in blood will be collected before the dose and 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 10, and 24 hours hours after the dose. Subjects will be allowed to leave the CRC after the 10 hour blood sample is collected and return the following day for the 24 hour sample.
2. Oseltamivir (Tamiflu®) 150 mg + Ethanol. In this phase, subjects will drink the same amount of orange juice over 15 minutes that will now have ethanol (alcohol) added. The amount of ethanol that will be added is calculated to achieve a blood alcohol concentration of 0.08 g/dl, which is considered to be legally intoxicated. Fifteen minutes after drinking the orange juice + ethanol, subjects will receive two (2) 75 mg capsules of oseltamivir with 5 ounces of water. Blood samples will be collected at the same times as above. An additional blood sample (1 teaspoonful) for determining the blood alcohol concentration will be collected 30 minutes after drinking the orange juice + ethanol.
3. Aspirin 650 mg. Subjects will drink orange juice (about 10 ounces although the amount may vary slightly based on your weight) over 15 minutes. Fifteen minutes after drinking the orange juice, they will take two (2) 325 mg aspirin tablets with 5 oz of water. Blood samples to determine the amount of aspirin in the blood will be collected before the aspirin dose and at 10, 20, and 30 minutes after the dose and at 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 5.0, 6.0, 7.0, and 8.0 hours after the dose.
4. Aspirin 650 mg + Ethanol. In this phase, subjects will drink the same amount of orange juice over 15 minutes that will now have ethanol (alcohol) added. The amount of ethanol that will be added is calculated to achieve a blood alcohol concentration of 0.08 g/dl, which is considered to be legally intoxicated. Fifteen minutes after drinking the orange juice + ethanol, subjects will take two (2) 325 mg aspirin tablets with 5 ounces of water. Blood samples (1 teaspoonful) to determine the amount of aspirin in the blood will be collected before the aspirin dose and at 10, 20, and 30 minutes after the dose and at 1.0, 1.5, 2.0, 2.5, 3.0, 4.0, 5.0, 6.0, 7.0, and 8.0 hours after the dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers ages 21-45 with no chronic medical or psychiatric conditions
* social ethanol drinker

Exclusion Criteria:

* allergy or hypersensitivity to oseltamivir or aspirin
* concomitant medication treatment (either prescription, over the counter, herbals, or supplements such as vitamins
* co-existing diseases affecting cardiovascular, hepatic, renal, pulmonary, hematologic, or gastrointestinal function
* platelet count < 100,000, hematocrit < 30
* chronic psychiatric disorder
* score >2 on the Michigan Alcohol Screening Test (MAST)
* naive to alcohol ingestion, have a family history of alcohol dependence, or history of adverse responses to alcohol
* women with known pregnancy, lactation, or not using and effective method of birth control (subjects taking oral contraceptives will be excluded)
* ingestion of alcohol or caffeine during the study
* participation in another drug study or blood donation within the preceding weeks.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2012-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve | Oseltamivir 0-24 hrs; Aspirin 0-8 hours
  For determining if ethanol inhibits hCE1 or hCE2, the primary pharmacokinetic parameter of interest will be the area under the plasma concentration-time curve from time zero to infinity (AUC0-∞) for oseltamivir phosphate and acetylsalicylic acid, respectively. Other pharmacokinetic parameters that will be characterized are maximum plasma concentration (Cmax), time to reach the maximum plasma concentration (tmax), and the elimination rate constant λz. This same pharmacokinetic analysis will also be applied to the oseltamivir carboxylate and salicylic acid metabolites. The change in the metabolite formation clearance (∆Clf) for each agent will be calculated as the ratio of the metabolite to parent AUC0-∞ when given with ethanol (inh) and alone (con) as follows: ΔClf = [AUCm/AUCp]inh/[AUCm/AUCp]con

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Parker, PharmD, Principal Investigator — University of Tennessee; Steven C Laizure, PharmD, Principal Investigator — University of Tennessee
Locations (1):
- University of Tennessee Health Science Center, Memphis, Tennessee, United States